CLINICAL TRIAL: NCT05675501
Title: Randomized, Double-Blind, Cross-Over, Vehicle Controlled Evaluation of Topical Encapsulated Benzoyl Peroxide on the Skin Microbiome and Skin Biophysical Properties
Brief Title: Evaluation of Topical Encapsulated Benzoyl Peroxide on the Skin Microbiome and Skin Biophysical Properties
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sol-Gel Technologies, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: SGT-54-08
Record Dates: First submitted 2022-12-01; First posted 2023-01-09 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Drug (Experimental): Daily Encapsulated Benzoyl Peroxide (E-BPO) Cream, for 8 weeks (period 1). Subjects will then switch treatments to the vehicle cream for a period of 4 weeks (period 2),
  Interventions: Drug: Encapsulated Benzoyl Peroxide Cream
- Vehicle (Placebo Comparator): Daily Vehicle Cream, for 8 weeks (period 1). Subjects will then switch treatments to the study drug encapsulated E-BPO for a period of 4 weeks (period 2),
  Interventions: Drug: Encapsulated Benzoyl Peroxide Cream

INTERVENTIONS:
Drug: Encapsulated Benzoyl Peroxide Cream — Subjects will use a "pea-size" amount for each area of the face

SUMMARY:
The overall objective of this study is to assess how the use of the drug may shift the skin microbiome and skin biophysical properties. Specifically, the study objectives were to assess the following:

* How the drug affects the skin microbiome compared with vehicle when applied once daily for 8 weeks in subjects with papulopustular rosacea.
* How the drug affects the skin physical properties compared with vehicle when applied once daily for 8 weeks in subjects with papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign an Institutional Review Board (IRB) approved written informed consent for this study.
* Male and female 18 years of age and older.
* Participants must have clinical diagnosis of moderate to severe rosacea.
* Have a minimum total of 15 and a maximum of 70 total inflammatory lesions (papules and/or pustules) including those present on the nose.
* Have 2 nodules or less.

Exclusion Criteria:

* Females, who are pregnant, breastfeeding, or planning a pregnancy within the period of their study participation or were found to have positive pregnancy test at Baseline or screening visits.
* Presence of more than 2 facial nodules or any nodule greater than 1 centimeter (cm).
* Current or past ocular rosacea (for example, conjunctivitis, blepharitis, or keratitis) of sufficient severity to require topical or systemic antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in skin microbiome diversity after 8-weeks of treatment compared to baseline | 8-weeks
  Facial microbiome sampling will be performed on-site by collecting follicular samples as well as utilizing facial swabs.
Change in transepidermal water loss after 8-weeks of treatment compared to baseline. | 8-weeks
  transepidermal water loss in g/m2/h
Change in stratum corneum hydration after 8-weeks of treatment compared to baseline. | 8-weeks
  stratum corneum water content (wt%)
Change in sebum excretion rate after 8-weeks of treatment compared to baseline. | 8-weeks
  sebum production in µg/cm2
Change in colorimeter test after 8-weeks of treatment compared to baseline. | 8-weeks
  facial L*a*b* values

SECONDARY OUTCOMES:
Change in skin microbiome diversity after 30 minutes, 1-week, 2-weeks and 4-weeks of treatment compared to baseline | 4-weeks
  Facial microbiome sampling will be performed on-site by collecting follicular samples as well as utilizing facial swabs.
Change in transepidermal water loss after 1-week, 2-weeks and 4-weeks of treatment compared to baseline. | 4-weeks
  transepidermal water loss in g/m2/h
Change in stratum corneum hydration after 1-week, 2-weeks and 4-weeks of treatment compared to baseline. | 4-weeks
  stratum corneum water content (wt%)
Change in sebum excretion rate after 1-week, 2-weeks and 4-weeks of treatment compared to baseline. | 4-weeks
  sebum production in µg/cm2
Change in colorimeter test after 1-week, 2-weeks and 4-weeks of treatment compared to baseline. | 4-weeks
  facial L*a*b* values

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research (ISSR), Sacramento, California, United States

REFERENCES:
- [Derived] Nong Y, Sugarman J, York JP, Levy-Hacham O, Nadora D, Mizrahi R, Galati A, Gallo RL, Sivamani RK. Effect of Topical Microencapsulated Benzoyl Peroxide on the Skin Microbiome in Rosacea: A Randomized, Double-Blind, Crossover, Vehicle-Controlled Clinical Trial. J Clin Aesthet Dermatol. 2024 Aug;17(8):19-26. PMID 39148964